CLINICAL TRIAL: NCT01829087
Title: Botulinum Toxin A to Treat Flexion Contracture After Total Knee Arthroplasty: A Double-Blinded Randomized Controlled Study
Brief Title: Botulinum Toxin A to Treat Flexion Contracture After Total Knee Arthroplasty
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Rothman Institute Orthopaedics (Other)
Collaborators: Sharpe-Strumia Research Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2012ES01
Record Dates: First submitted 2013-04-08; First posted 2013-04-11 (Estimated); Last update posted 2013-12-13 (Estimated); Status verified 2013-12

CONDITIONS: Flexion Contracture Following Total Knee Replacement
MeSH Terms: interventions — Botulinum Toxins, Type A

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Botox injection (Experimental)
  Interventions: Drug: Botox
- Control (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Botox
  Arms: Botox injection
Drug: placebo
  Arms: Control

SUMMARY:
The goal of this research project is to evaluate injections of botulinum toxin A (Botox) as the treatment for knee flexion contracture after total knee arthroplasty (TKA). The current treatment for patients who do not achieve full extension of the knee (flexion contracture) after TKA consists of an aggressive physical therapy program, home stretching program, and the use of an extension orthosis (brace). Many patients do not tolerate wearing these braces. This initial project is designed to use injections of Botox as an adjunct to the standard current treatment and evaluate its efficacy. It is our hypothesis that a single injection into the hamstrings in addition to routine postoperative rehabilitation will result in improved knee extension and this improvement in function should endure without further treatment.

ELIGIBILITY:
Inclusion Criteria:

* Subject is at least 18 years of age
* Subject had a total knee replacement or total knee replacement revision surgery performed at Main Line hospitals such as Bryn Mawr Hospital, Lankenau Hospital, and Riddle Hospital
* Subject is measured to have at least 10 degree flexion contracture of the operative knee four to six weeks following surgery
* Subject has the willingness to complete scheduled follow up evaluations as described in the informed consent

Exclusion Criteria:

* Subject is currently involved in another study or has received investigational product or treatment within the last 30 days
* Subject is a prisoner
* Subject is anticipated to be non-compliant
* Subject is known to be pregnant
* Subject is mentally incompetent or unable to understand what participation in the study entails
* The subject has a known sensitivity or allergic reaction to Botulinum Toxin A and albumin
* The subject is unwilling or unable to give consent or to comply with the follow up program

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2012-08; Primary Completion 2014-08 (Estimated)

PRIMARY OUTCOMES:
Range of Motion: knee | 1 year

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Rothman Institute, Bryn Mawr, Pennsylvania
  - Rothman Institute, Lankenau, Pennsylvania